CLINICAL TRIAL: NCT02249923
Title: Pediatric Pulmonary Hypertension Network (PPHNet) Informatics Registry
Acronym: PPHNet
Status: Recruiting | Type: Observational
Sponsor: New York Medical College (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-0018; U01HL121518 (NIH); NOPRODPUH4017 (Other Grant/Funding Number: Department of Education)
Record Dates: First submitted 2014-09-10; First posted 2014-09-26 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Vascular Disease; Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension (PAH); Pulmonary Vascular Disease (PVD); Registry; Pediatric
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pulmonary Arterial Hypertension

SUMMARY:
Patients are being asked to be in this research study because medical researchers hope that by gathering information about a large number of children with pulmonary hypertension over time, their understanding of the disease process will increase and lead to better treatment. Investigators believe that pulmonary hypertension in children is different than pulmonary hypertension in adults and this study will help us understand those differences.

DETAILED DESCRIPTION:
Pulmonary Hypertension (PH) is a syndrome characterized by vasoconstriction and abnormal growth and function of endothelial and smooth muscle cells and other components within the pulmonary vessels, which leads to elevation of the pulmonary artery pressure. PH may be idiopathic (primary) without any known cause. Some cases of PH are familial. PH may also be secondary to a specific disease process such as portal hypertension, congenital heart disease, chronic lung disease, thromboembolic disease, connective tissue disease, human immunodeficiency virus (HIV), and use of anorexigens. Left untreated, PH is often progressive and fatal. There is no cure for PH. Therapy focuses upon treatment of secondary causes if present, and reduction of the pulmonary artery pressure through medical therapy. There have been many new developments within the past few years in the management of patients with PH. While there is no cure for PH early detection and treatment are important for survival of patients. Limited data is available that describes the etiologies, clinical course and prognosis of pediatric pulmonary hypertension.

Objectives

Aim 1: Clinical Research

1. To provide a mechanism to store information about newborns, infants and children with PH;
2. To determine the incidence and natural history of the various etiologies of pediatric PH;
3. To define the investigator current diagnostic and therapeutic approaches to the diverse conditions associated with pediatric PH;
4. To determine the response of children with PH to chronic therapies.

Aim 2: Research Infrastructure To create a robust scalable data architecture, to combine traditional registry data, electronic Health Record (EHR), and PRO (Patient Reported Outcome) data in a single resource.

Aim 3: Informatics Address three classes of unanswered questions crucial for the characterization and management of PH, comparing the information value of registry vs. EHR vs. fused data across registry/EHR/PROs, in the domains of spectrum of PH comorbidities, PH indicators and endpoints of morbidity and mortality, and response to therapies in PH.

Aim 4: Risk Stratification To validate the Pediatric Risk Score model using an independent patient cohort, obtained by enrichment of the PPHNet Registry with phenotypic data collection from a newly enrolled cohort of 500 patients (Collaborative substudy with Johnson & Johnson- "Children Are Not Small Adults: Validation of the Pediatric Pulmonary Hypertension Risk Score")

ELIGIBILITY:
Inclusion Criteria:

* The subject's age of onset of pulmonary hypertension must be prior to age 18 years
* The person providing consent must be able to read either Spanish or English.
* The subject (and/or parent/legal guardian) must be able to provide informed consent

Exclusion Criteria:

* Diagnosed with pulmonary hypertension after age 18
* Refusal to sign informed consent

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pulmonary Hypertension (PH) is a syndrome characterized by vasoconstriction and abnormal growth and function of endothelial and smooth muscle cells and other components within the pulmonary vessels, which leads to elevation of the pulmonary artery pressure. PH may be idiopathic (primary) without any known cause. Some cases of PH are familial. PH may also be secondary to a specific disease process such as portal hypertension, congenital heart disease, chronic lung disease, thromboembolic disease, connective tissue disease, HIV, and use of anorexigens.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2014-10; Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Time to clinical worsening | 12 months
  Time to clinical worsening for death, cardiac transplant, atrial septostomy, or Potts shunt.

SECONDARY OUTCOMES:
Escalation of Pulmonary Hypertension Therapy | 36 months
  The addition of patients baseline medication therapy, this can include going from mono therapy to dual therapy, or dual therapy to triple therapy
Right Heart Failure | 36 months
  Elevated Right atrial pressure greater than 10 by right heart catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Abman, MD, Principal Investigator — Children's Hospital Colorado; David D Ivy, MD, Principal Investigator — Children's Hospital Colorado; Kenneth D Mandl, MD, Principal Investigator — Boston Children's Hospital, Harvard School of Medicine; Roberta Keller, MD, Principal Investigator — University California San Francisco; Rachel Hopper, MD, Principal Investigator — Stanford University; Angela Bates, MD, Principal Investigator — University of Alberta Edmonton; Catherine Avitabile, MD, Principal Investigator — Children's Hospital of Philadelphia; Mary Mullen, MD, Principal Investigator — Boston Children's Hospital; Eric Austin, MD, Principal Investigator — Vanderbilt University Medical Center; Marc Natter, MD, Principal Investigator — Boston Children's Hospital; Usha Krishnan, MD, Principal Investigator — Columbia University; Lynn A Sleeper, ScD, Principal Investigator — Boston Children's Hospital; Erika Rosenzweig, MD, Principal Investigator — Maria Fareri Children's Hospital at WMC Health/Westchester Medical Center; Jenny Schramm, MD, Principal Investigator — Johns Hopkins University; Lewis Romer, MD, Principal Investigator — Johns Hopkins University; Grace Freire, MD, Principal Investigator — Johns Hopkins All Children's Heart Institute; Stephanie Handler, MD, Principal Investigator — Children's Hospital Wisconsin; Nidhy Varghese, MD, Principal Investigator — Baylor College of Medicine; Russel Hirsch, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Delphine Yung, MD, Principal Investigator — Seattle Children's Hospital
Locations (14):
- United States (13):
  - Stanford University Medical Center, Palo Alto, California
  - University California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Johns Hopkins All Children's Heart Institute, St. Petersburg, Florida
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Maria Fareri Children's Hospital at WMC Health/Westchester Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- University of Alberta Edmonton, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geva A, Gronsbell JL, Cai T, Cai T, Murphy SN, Lyons JC, Heinz MM, Natter MD, Patibandla N, Bickel J, Mullen MP, Mandl KD; Pediatric Pulmonary Hypertension Network and National Heart, Lung, and Blood Institute Pediatric Pulmonary Vascular Disease Outcomes Bioinformatics Clinical Coordinating Center Investigators. A Computable Phenotype Improves Cohort Ascertainment in a Pediatric Pulmonary Hypertension Registry. J Pediatr. 2017 Sep;188:224-231.e5. doi: 10.1016/j.jpeds.2017.05.037. Epub 2017 Jun 16. PMID 28625502
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/34140292/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/35049414/